CLINICAL TRIAL: NCT06181058
Title: The Effect of the Escape Room Game on Students' Academic Self-Efficacy and Critical Thinking: An Oncology Nursing Course Example
Brief Title: Escape Room Game in Oncology Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuğçe Türten Kaymaz, asisstant professor, Ankara Yildirim Beyazıt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AnkaraYBU-SBF-TTK-01
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Oncology; Education
Keywords: game; self efficacy; thinking; student; oncology nursing; education
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The participant list will be uploaded to a program and teams of 6-8 people will be formed with random names. The participant list will be uploaded to a program and teams of 6-8 people will be formed with random names. Each team will play the escape game.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- escape room game (Experimental): The participant list will be uploaded to a program and teams of 6-8 people will be formed with random names. The participant list will be uploaded to a program and teams of 6-8 people will be formed with random names. Each team will play the escape game.
  Participants will be informed about the game. He/she will be asked to solve puzzles within the framework of an oncology patient scenario. There will be a debriefing session at the end of the escape game.
  Participants will be informed with a scenario containing the story of an oncology patient, and puzzles-riddles related to the case will be given within the game. They will get a letter when they solve each riddle and complete the game by solving the password.
  Interventions: Behavioral: escape room game

INTERVENTIONS:
Behavioral: escape room game — Participants will be informed about the game (15 minutes). They will complete the game by solving puzzles within the framework of the oncology patient scenario (approximately 30 minutes). There will be a debriefing session at the end of the escape game (15 minutes).

SUMMARY:
This research will be conducted to evaluate the effect of the escape room game activity applied to nursing students taking oncology nursing courses on their academic self-efficacy and critical thinking motivation.

DETAILED DESCRIPTION:
Considering the characteristics of cancer patients and the complexity of care, it is essential to include a separate oncology nursing course in the education curriculum to increase the qualifications of nursing students. During undergraduate nursing education, clinical practices for care in oncological diseases are limited. New approaches are needed that will contribute to increasing the effectiveness of the educational processes of nursing students. Escape room game-based educational approaches, which have begun to be used in nursing education in recent years, are presented as an example of this situation. Escape games are defined as a type of student-centered activity designed to improve students' learning and skills in professional development programs. The main purpose of using escape games in nursing education is to create practice environments where students will gain clinical decision-making competence in order to provide safe and qualified patient care services. This research was designed to determine the effect of the escape room game applied to students taking oncology nursing courses on their academic self-efficacy and critical thinking motivation.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in the Oncology Nursing course and volunteering to participate in the study

Exclusion Criteria:

* Not completing the game during the escape room game and/or filling in the scales and forms incompletely

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Academic Self-Efficacy Scale | First assessment; after the pre-briefing, immediately before the game. Second assessment; immediately after the debriefing, approximately 15 minute after the game.
  The scale consists of 4 sub-dimensions and 14 items. An increase in the score obtained indicates that the student's academic self-efficacy also increases.

SECONDARY OUTCOMES:
Critical Thinking Motivation Scale | First assessment; after the pre-briefing, immediately before the game. Second assessment; immediately after the debriefing, approximately 15 minute after the game .
  This scale was developed to provide information about motivation for a specific critical thinking task. The scale consists of 19 Likert-type items ranging from 1 to 6 (1 = "I Strongly Disagree" and 6 = "I Strongly Agree"). The scale consists of two main sub-dimensions named "expectation" and "value". An increase in the score obtained from the scale indicates that the student's critical thinking motivation has increased.
Game-X Scale | Immediately after the debriefing, approximately 15 minute after the game.
  The scale was developed in 2018 to evaluate game experiences. In this scale, factors covering six dimensions namely absorption, enjoyment, activation, creative thinking, absence of negativity and dominance. The scale consists of 27 questions and 6 sub-dimensions. The scale is Likert type and responses are scored between 1 (never) and 5 (always). An increase in the score obtained indicates that the gaming experience is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe Türten Kaymaz, PhD, Principal Investigator — Ankara Yildirim Beyazıt University; Betül Çakmak, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No